CLINICAL TRIAL: NCT04446039
Title: Comparison of Antidepressants in the Real-World: Retrospective Cohort Study Using Big Data
Brief Title: Non-interventional, Retrospective Cohort Study to Explore Antidepressant Treatment in Korea
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B2061147; CAR-BIG Study (Other: Alias Study Number)
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; Paroxetine; Fluoxetine; Mirtazapine; Duloxetine Hydrochloride; Sertraline; Venlafaxine Hydrochloride; tianeptine; Vortioxetine; Desvenlafaxine Succinate; Bupropion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (11):
- 1. Escitalopram Cohort
  Interventions: Drug: Escitalopram
- 2. Paroxetine Cohort
  Interventions: Drug: Paroxetine
- 3. Fluoxetine Cohort
  Interventions: Drug: Fluoxetine
- 4. Mirtazapine Cohort
  Interventions: Drug: Mirtazapine
- 5. Duloxetine Cohort
  Interventions: Drug: Duloxetine
- 6. Sertraline Cohort
  Interventions: Drug: Sertraline
- 7. Venlafaxine Cohort
  Interventions: Drug: Venlafaxine
- 8. Tianeptine Cohort
  Interventions: Drug: Tianeptine
- 9. Vortioxetine Cohort
  Interventions: Drug: Vortioxetine
- 10. Desvenlafaxine Cohort
  Interventions: Drug: Desvenlafaxine
- 11. Bupropion Cohort
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Escitalopram — Treatment for depression
  Groups: 1. Escitalopram Cohort
Drug: Paroxetine — Treatment for depression
  Groups: 2. Paroxetine Cohort
Drug: Fluoxetine — Treatment for depression
  Groups: 3. Fluoxetine Cohort
Drug: Mirtazapine — Treatment for depression
  Groups: 4. Mirtazapine Cohort
Drug: Duloxetine — Treatment for depression
  Groups: 5. Duloxetine Cohort
Drug: Sertraline — Treatment for depression
  Groups: 6. Sertraline Cohort
Drug: Venlafaxine — Treatment for depression
  Groups: 7. Venlafaxine Cohort
Drug: Tianeptine — Treatment for depression
  Groups: 8. Tianeptine Cohort
Drug: Vortioxetine — Treatment for depression
  Groups: 9. Vortioxetine Cohort
Drug: Desvenlafaxine — Treatment for depression
  Groups: 10. Desvenlafaxine Cohort
Drug: Bupropion — Treatment for depression
  Groups: 11. Bupropion Cohort

SUMMARY:
The primary purpose of this study is to investigate medication utilization pattern and risk of adverse outcomes among commonly used antidepressants by using nationwide claims database, in order to assess overall clinical benefit of antidepressant therapy in real-world practice.

DETAILED DESCRIPTION:
While there are many antidepressants from which physicians can select based on efficacy and tolerability profile, evidence on effectiveness and safety outcomes of new antidepressants in real clinical practice among Korean MDD population is limited.

Hence, this study will explore the following primary, secondary objectives using national health insurance database :

1. Explore baseline characteristics and drug utilization patterns of 11 commonly used antidepressant therapy during 90 days of acute treatment phase
2. Explore drug utilization patterns such as therapy changes, medication compliance and recurrence relationship, and risk of adverse outcomes during maintenance phase
3. Choice of antidepressants and drug utilization patterns in patients with various comorbidities
4. The relationship of non-pharmacologic treatment and discontinuation, medication compliance
5. Choice of antidepressants by non-psychiatric specialty

ELIGIBILITY:
Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Patients aged 18 years or older on the index date
2. Patients who had at least one inpatient claim or two outpatient claims in the intake period with any of the following diagnosis codes F06.3 Organic mood [affective] disorders F32* Depressive episode F33* Recurrent depressive disorder F34.1 Neurotic depression F38.1 Other recurrent mood [affective] disorder F41.2 Mixed anxiety and depressive disorder
3. Patients prescribed any of the following antidepressant during intake period (from January 1, 2017 to June 30, 2018)

Exclusion Criteria

Patients meeting any of the following criteria will not be included in the study:

1. Patients with a claim of diagnosis codes in Table 1 during the 12 month pre-index period
2. Patients with a claim of prescription in Table 2 during the 12 month pre-index period
3. Patient who had a claim as a beneficiary of Medical Aid program (Korean Medicaid program with free or minimum copay)
4. Patients who are hospitalized at the index date
5. Patients who are under hospice care (procedure codes WG*-WO*)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who newly initiated antidepressant therapies between Jan 01, 2017 to Jun 30, 2018 in the National Health Insurance Service (NHIS) database
Sampling Method: Probability Sample
Enrollment: 370212 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B2061147

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who initiated antidepressants between 01-Jan-2018 to 30-Jun-2019 in Health Insurance Review and Assessment (HIRA) service database were observed in this retrospective study. Index date was first prescription date of study drugs during intake period (01-Jan-2018 to 31-Dec-2019). Acute phase was initial 90 days of treatment period and maintenance phase was from 91 to 180 days of treatment. Participants were followed up until 31-Dec-2020.
Pre-assignment Details: A total of 370212 participants were included in the study.
Groups:
- Participants With Antidepressant Therapy: Participants who initiated antidepressant therapy (escitalopram, paroxetine, fluoxetine, mirtazapine, duloxetine, sertraline, venlafaxine, tianeptine, vortioxetine, desvenlafaxine and bupropion) between 01-Jan-2018 to 30-Jun-2019 in the HIRA database were included and observed.
Period: Overall Study
Arm/Group | Participants With Antidepressant Therapy
Started | 370212
Completed | 370212
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included participants who had newly initiated antidepressant therapies between 01-Jan-2018, to 30-Jun-2019, in the HIRA database.
Arm/Group | Participants With Antidepressant Therapy
Number analyzed (Participants) | 370212
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.51 (15.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 223994
  Male | 146218
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Medication Possession Ratio (MPR) During First 180 Days of Treatment
Description: MPR= Days of medication possession from the prescriptions filled in the 180 days divided by (180 days plus + extra days of drug supply from the last prescription fill during the 180 days). MPR by each index drug including escitalopram, paroxetine, fluoxetine, mirtazapine, duloxetine, sertraline, venlafaxine, tianeptine, vortioxetine, desvenlafaxine and bupropion is reported in this outcome measure. Index date was first prescription date of study drugs during intake period.
Time Frame: From index date (anytime between 01-Jan-2018 to 31-Dec-2019) up to 180 days of treatment (data collected and observed retrospectively)
Population: FAS included participants who had newly initiated antidepressant therapies between 01-Jan-2018 to 30-Jun-2019, in the HIRA database. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Participants With Antidepressant Therapy
Number analyzed (Participants) | 370212
Ratio
  Escitalopram: number analyzed (Participants) | 178740
  Escitalopram | 0.47 (0.35)
  Paroxetine: number analyzed (Participants) | 37154
  Paroxetine | 0.49 (0.36)
  Fluoxetine: number analyzed (Participants) | 44,069
  Fluoxetine | 0.46 (0.34)
  Sertraline: number analyzed (Participants) | 31,285
  Sertraline | 0.48 (0.36)
  Duloxetine: number analyzed (Participants) | 8,449
  Duloxetine | 0.47 (0.36)
  Venlafaxine: number analyzed (Participants) | 7,726
  Venlafaxine | 0.50 (0.36)
  Desvenlafaxine: number analyzed (Participants) | 4,637
  Desvenlafaxine | 0.53 (0.36)
  Mirtazapine: number analyzed (Participants) | 11,414
  Mirtazapine | 0.47 (0.36)
  Tianeptine: number analyzed (Participants) | 24,536
  Tianeptine | 0.39 (0.33)
  Vortioxetine: number analyzed (Participants) | 14,504
  Vortioxetine | 0.50 (0.35)
  Bupropion: number analyzed (Participants) | 7,698
  Bupropion | 0.45 (0.34)

2. Primary Outcome: Persistence During First 180 Days of Treatment
Description: Persistence was defined as the average length of treatment on the index drugs (escitalopram, paroxetine, fluoxetine, mirtazapine, duloxetine, sertraline, venlafaxine, tianeptine, vortioxetine, desvenlafaxine and bupropion), allowing 14-day permissible gap. Index date was first prescription date of study drugs during intake period.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Participants With Antidepressant Therapy
Number analyzed (Participants) | 370212
Days
  Escitalopram: number analyzed (Participants) | 178,740
  Escitalopram | 76.11 (67.04)
  Paroxetine: number analyzed (Participants) | 37,154
  Paroxetine | 79.83 (68.43)
  Fluoxetine: number analyzed (Participants) | 44,069
  Fluoxetine | 74.17 (65.32)
  Sertraline: number analyzed (Participants) | 31,285
  Sertraline | 77.34 (67.64)
  Duloxetine: number analyzed (Participants) | 8,449
  Duloxetine | 71.66 (67.64)
  Venlafaxine: number analyzed (Participants) | 7,726
  Venlafaxine | 79.80 (68.79)
  Desvenlafaxine: number analyzed (Participants) | 4,637
  Desvenlafaxine | 87.13 (68.81)
  Mirtazapine: number analyzed (Participants) | 11,414
  Mirtazapine | 73.12 (66.78)
  Tianeptine: number analyzed (Participants) | 24,536
  Tianeptine | 54.48 (60.14)
  Vortioxetine: number analyzed (Participants) | 14,504
  Vortioxetine | 81.44 (66.50)
  Bupropion: number analyzed (Participants) | 7,698
  Bupropion | 71.96 (63.82)

3. Primary Outcome: Percentage of Participants Who Discontinued Treatment in the First 90 Days From the Index Date
Description: Percentage of participants who discontinued the treatment in first 90 days from the index date is reported in this outcome measure. Index date was the first prescription date of study treatment during the intake period.
Time Frame: From the index date (anytime between 01-Jan-2018 to 30-Jun-2019) up to 90 days of treatment (data collected and observed retrospectively)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Antidepressant Therapy
Number analyzed (Participants) | 370212
Percentage of participants
  Escitalopram: number analyzed (Participants) | 178740
  Escitalopram | 14.82
  Paroxetine: number analyzed (Participants) | 37154
  Paroxetine | 15.16
  Fluoxetine: number analyzed (Participants) | 44069
  Fluoxetine | 15.14
  Sertraline: number analyzed (Participants) | 31285
  Sertraline | 14.87
  Duloxetine: number analyzed (Participants) | 8449
  Duloxetine | 17.04
  Venlafaxine: number analyzed (Participants) | 7726
  Venlafaxine | 14.04
  Desvenlafaxine: number analyzed (Participants) | 4637
  Desvenlafaxine | 12.81
  Mirtazapine: number analyzed (Participants) | 11414
  Mirtazapine | 15.21
  Tianeptine: number analyzed (Participants) | 24536
  Tianeptine | 22.27
  Vortioxetine: number analyzed (Participants) | 14504
  Vortioxetine | 12.94
  Bupropion: number analyzed (Participants) | 7698
  Bupropion | 14.34

4. Primary Outcome: Percentage of Participants Who Adhered to Treatment Measured by MPR (More Than or Equal to [>=] 75 Percent [%])
Description: Adherence was defined when MPR >= 75%. MPR = (Days of medication possession from the prescriptions filled in the 180 days) / (180 days + extra days of drug supply from the last prescription fill during the 180 days. Index date was the first prescription date of study drugs during the intake period.
Time Frame: From the index date (anytime between 01-Jan-2018 to 30-Jun-2019) up to 180 days of treatment (data collected and observed retrospectively)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Antidepressant Therapy
Number analyzed (Participants) | 370212
Percentage of participants
  Escitalopram: number analyzed (Participants) | 178740
  Escitalopram | 30.31
  Paroxetine: number analyzed (Participants) | 37154
  Paroxetine | 33.18
  Fluoxetine: number analyzed (Participants) | 44069
  Fluoxetine | 27.92
  Sertraline: number analyzed (Participants) | 31285
  Sertraline | 31.48
  Duloxetine: number analyzed (Participants) | 8449
  Duloxetine | 30.73
  Venlafaxine: number analyzed (Participants) | 7726
  Venlafaxine | 33.39
  Desvenlafaxine: number analyzed (Participants) | 4637
  Desvenlafaxine | 37.20
  Mirtazapine: number analyzed (Participants) | 11414
  Mirtazapine | 30.32
  Tianeptine: number analyzed (Participants) | 24536
  Tianeptine | 20.75
  Vortioxetine: number analyzed (Participants) | 14504
  Vortioxetine | 32.51
  Bupropion: number analyzed (Participants) | 7698
  Bupropion | 27.16

5. Primary Outcome: Percentage of Participants Experiencing Recurrence During the Acute Treatment Phase
Description: Recurrence during the acute treatment phase was defined as either one of the following: 1) Inpatient episode with a diagnosis code. 2) Inpatient episodes via the department of psychiatry or emergency medicine. 3) Inpatient episode via nursing hospital. 4) Emergency room visit with a diagnosis code. 5) Suicide attempt. Acute phase considered as the first 90-day period starting from the index date. Index date was the first prescription date of study treatment during the intake period. Diagnosis codes used for inclusion were: F06.3-Organic mood(affective) disorders, F32*- Depressive episode, F33*- Recurrent depressive disorder, F34.1- Neurotic depression, F38.1- Other recurrent mood(affective) disorders, F41.2- Mixed anxiety and depressive disorder.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Antidepressant Therapy
Number analyzed (Participants) | 370212
Percentage of participants
  Escitalopram: number analyzed (Participants) | 178740
  Escitalopram | 16.42
  Paroxetine: number analyzed (Participants) | 37154
  Paroxetine | 17.84
  Fluoxetine: number analyzed (Participants) | 44069
  Fluoxetine | 15.64
  Sertraline: number analyzed (Participants) | 31285
  Sertraline | 16.73
  Duloxetine: number analyzed (Participants) | 8449
  Duloxetine | 17.97
  Venlafaxine: number analyzed (Participants) | 7726
  Venlafaxine | 17.73
  Desvenlafaxine: number analyzed (Participants) | 4637
  Desvenlafaxine | 20.85
  Mirtazapine: number analyzed (Participants) | 11414
  Mirtazapine | 19.51
  Tianeptine: number analyzed (Participants) | 24536
  Tianeptine | 16.34
  Vortioxetine: number analyzed (Participants) | 14504
  Vortioxetine | 17.62
  Bupropion: number analyzed (Participants) | 7698
  Bupropion | 16.13

6. Primary Outcome: Percentage of Participants Experiencing Recurrence After the Acute Treatment Phase
Description: Recurrence was defined as either one of the following: 1) Inpatient episode with a diagnosis code. 2) Inpatient episodes via the department of psychiatry or emergency medicine. 3) Inpatient episode via nursing hospital. 4) Emergency room visit with a diagnosis code. 5) Suicide attempt; antidepressant prescription after 30 days of drug holiday. Acute phase considered as the first 90-day period starting from the index date. Index date was the first prescription date of study treatment during the intake period.
Time Frame: From day 91 to day 180 from the index date (anytime between 01-Jan-2018 to 30-Jun-2019) (data collected and observed retrospectively)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Antidepressant Therapy
Number analyzed (Participants) | 370212
Percentage of participants
  Escitalopram: number analyzed (Participants) | 178740
  Escitalopram | 22.71
  Paroxetine: number analyzed (Participants) | 37154
  Paroxetine | 23.58
  Fluoxetine: number analyzed (Participants) | 44069
  Fluoxetine | 23.74
  Sertraline: number analyzed (Participants) | 31285
  Sertraline | 22.91
  Duloxetine: number analyzed (Participants) | 8449
  Duloxetine | 25.48
  Venlafaxine: number analyzed (Participants) | 7726
  Venlafaxine | 23.36
  Desvenlafaxine: number analyzed (Participants) | 4637
  Desvenlafaxine | 23.81
  Mirtazapine: number analyzed (Participants) | 11414
  Mirtazapine | 24.64
  Tianeptine: number analyzed (Participants) | 24536
  Tianeptine | 27.80
  Vortioxetine: number analyzed (Participants) | 14504
  Vortioxetine | 22
  Bupropion: number analyzed (Participants) | 7698
  Bupropion | 21.85

7. Primary Outcome: Percentage of Participants With Adverse Events (AE) Within Maintenance Phase of Treatment
Description: An AE was any untoward medical occurrence that did not necessarily have a causal relationship with study treatment. Maintenance phase was during the second 90-day period (91 to 180 days) starting from the index date. Index date was the first prescription date of study treatment during the intake period. Index date was the first prescription date of study treatment during the intake period.
Time Frame: From 91 up to 180 days of treatment from index date (anytime between 01-Jan-2018 to 30-Jun-2019) (data collected and observed retrospectively)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Participants With Antidepressant Therapy
Number analyzed (Participants) | 370212
Percentage of Participants
  Escitalopram: number analyzed (Participants) | 178740
  Escitalopram | 6.08
  Paroxetine: number analyzed (Participants) | 37154
  Paroxetine | 6.44
  Fluoxetine: number analyzed (Participants) | 44069
  Fluoxetine | 4.29
  Sertraline: number analyzed (Participants) | 31285
  Sertraline | 6.09
  Duloxetine: number analyzed (Participants) | 8449
  Duloxetine | 9.59
  Venlafaxine: number analyzed (Participants) | 7726
  Venlafaxine | 6.48
  Desvenlafaxine: number analyzed (Participants) | 4637
  Desvenlafaxine | 7.50
  Mirtazapine: number analyzed (Participants) | 11414
  Mirtazapine | 10.36
  Tianeptine: number analyzed (Participants) | 24536
  Tianeptine | 8.66
  Vortioxetine: number analyzed (Participants) | 14504
  Vortioxetine | 5.34
  Bupropion: number analyzed (Participants) | 7698
  Bupropion | 4.68

8. Primary Outcome: Percentage of Prescriptions for Commonly Used Antidepressants in Acute Treatment Phase
Description: Percentage of prescriptions for commonly used antidepressants in acute treatment phase were assessed. Acute treatment phase was during the first 90-day period starting from the index date. Index date was the first prescription date of study treatment during the intake period.
Time Frame: as for outcome 3
Population: FAS included participants who had newly initiated antidepressant therapies between 01-Jan-2018 to 30-Jun-2019, in the HIRA database.
Measure: Number; unit: Percentage of prescriptions
Units Other Than Participants: Prescriptions for antidepressants
Arm/Group | Participants With Antidepressant Therapy
Number analyzed (Participants) | 370212
Number analyzed (Prescriptions for antidepressants) | 2574691
Percentage of prescriptions
  Escitalopram | 44.19
  Paroxetine | 10.1
  Fluoxetine | 12.15
  Sertraline | 8.89
  Duloxetine | 2.3
  Venlafaxine | 3.21
  Desvenlafaxine | 1.75
  Mirtazapine | 4.1
  Tianeptine | 5.52
  Vortioxetine | 4.81
  Bupropion | 2.88

9. Primary Outcome: Average Daily Dosage at Index Date
Description: Index date was the first prescription date of study treatment during the intake period.
Time Frame: At index date (anytime between 01-Jan-2018 to 30-Jun-2019) (data collected and observed retrospectively)
Population: FAS included participants who had newly initiated antidepressant therapies between 01-Jan-2018, to 30-Jun-2019, in the HIRA database. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Milligrams per day
Arm/Group | Participants With Antidepressant Therapy
Number analyzed (Participants) | 370212
Milligrams per day
  Escitalopram: number analyzed (Participants) | 178740
  Escitalopram | 6.34 (3.23)
  Paroxetine: number analyzed (Participants) | 37154
  Paroxetine | 13.01 (5.50)
  Fluoxetine: number analyzed (Participants) | 44069
  Fluoxetine | 16.30 (8.55)
  Sertraline: number analyzed (Participants) | 31285
  Sertraline | 38.75 (19.56)
  Duloxetine: number analyzed (Participants) | 8449
  Duloxetine | 34.80 (12.91)
  Venlafaxine: number analyzed (Participants) | 7726
  Venlafaxine | 54.11 (29.12)
  Desvenlafaxine: number analyzed (Participants) | 4637
  Desvenlafaxine | 51.91 (11.32)
  Mirtazapine: number analyzed (Participants) | 11414
  Mirtazapine | 8.71 (5.56)
  Tianeptine: number analyzed (Participants) | 24536
  Tianeptine | 24.28 (9.24)
  Vortioxetine: number analyzed (Participants) | 14504
  Vortioxetine | 6.03 (2.62)
  Bupropion: number analyzed (Participants) | 7698
  Bupropion | 152.97 (53.43)

10. Primary Outcome: Average Daily Dosage During the Acute Treatment Phase
Description: Acute treatment phase was during the first 90-day period starting from the index date.
Time Frame: as for outcome 3
Population: FAS included participants who had newly initiated antidepressant therapies between 01-Jan-2018 to 30-Jun-2019, in the HIRA database. Here, 'Overall Number of Participants Analyzed' signifies number of participants who were treated with monotherapy and 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Milligrams per day
Arm/Group | Participants With Antidepressant Therapy
Number analyzed (Participants) | 278422
Milligrams per day
  Escitalopram: number analyzed (Participants) | 141056
  Escitalopram | 7.94 (4.13)
  Paroxetine: number analyzed (Participants) | 27160
  Paroxetine | 15.27 (7.48)
  Fluoxetine: number analyzed (Participants) | 32897
  Fluoxetine | 19.07 (10.34)
  Sertraline: number analyzed (Participants) | 23262
  Sertraline | 49.91 (30.24)
  Duloxetine: number analyzed (Participants) | 5822
  Duloxetine | 37.51 (16.62)
  Venlafaxine: number analyzed (Participants) | 5221
  Venlafaxine | 69.12 (39.98)
  Desvenlafaxine: number analyzed (Participants) | 3179
  Desvenlafaxine | 63.22 (26.91)
  Mirtazapine: number analyzed (Participants) | 8129
  Mirtazapine | 10.46 (7.15)
  Tianeptine: number analyzed (Participants) | 16030
  Tianeptine | 21.71 (9.85)
  Vortioxetine: number analyzed (Participants) | 10520
  Vortioxetine | 8.26 (3.95)
  Bupropion: number analyzed (Participants) | 5146
  Bupropion | 162.75 (67.75)

11. Other Pre Specified Outcome: Percentage of Participants on Monotherapy, Combination Therapy, Augmentation Therapy During Acute Treatment Phase
Description: Percentage of participants who received monotherapy, combination therapy and augmentation therapy during 90 days of treatment were assessed in this outcome measure. Acute treatment phase was during initial 90 days from the index date.
Time Frame: as for outcome 3
Population: FAS included participants who had newly initiated antidepressant therapies between 01-Jan-2018 to 30-Jun-2019, in the HIRA database. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified rows. One participant was evaluable for more than one row.
Measure: Number; unit: Percentage of Participants
Arm/Group | Participants With Antidepressant Therapy
Number analyzed (Participants) | 278422
Percentage of Participants
  Monotherapy: Escitalopram: number analyzed (Participants) | 178740
  Monotherapy: Escitalopram | 78.92
  Combination: Escitalopram: number analyzed (Participants) | 178740
  Combination: Escitalopram | 8.91
  Augmentation therapy: escitalopram: number analyzed (Participants) | 178740
  Augmentation therapy: escitalopram | 14.01
  Monotherapy: Paroxetine: number analyzed (Participants) | 37154
  Monotherapy: Paroxetine | 73.10
  Combination: Paroxetine: number analyzed (Participants) | 37154
  Combination: Paroxetine | 10.91
  Augmentation therapy: paroxetine: number analyzed (Participants) | 37154
  Augmentation therapy: paroxetine | 15.18
  Monotherapy: Fluoxetine: number analyzed (Participants) | 44069
  Monotherapy: Fluoxetine | 74.65
  Combination: Fluoxetine: number analyzed (Participants) | 44069
  Combination: Fluoxetine | 10.08
  Augmentation therapy: fluoxetine: number analyzed (Participants) | 44069
  Augmentation therapy: fluoxetine | 13.52
  Monotherapy: Sertraline: number analyzed (Participants) | 31285
  Monotherapy: Sertraline | 74.36
  Combination: Sertraline: number analyzed (Participants) | 31285
  Combination: Sertraline | 9.37
  Augmentation therapy: sertraline: number analyzed (Participants) | 31285
  Augmentation therapy: sertraline | 14.16
  Monotherapy: Duloxetine: number analyzed (Participants) | 8449
  Monotherapy: Duloxetine | 68.91
  Combination: Duloxetine: number analyzed (Participants) | 8449
  Combination: Duloxetine | 12.53
  Augmentation therapy: duloxetine: number analyzed (Participants) | 8449
  Augmentation therapy: duloxetine | 14.31
  Monotherapy: Venlafaxine: number analyzed (Participants) | 7726
  Monotherapy: Venlafaxine | 67.58
  Combination: Venlafaxine: number analyzed (Participants) | 7726
  Combination: Venlafaxine | 13.11
  Augmentation therapy: venlafaxine: number analyzed (Participants) | 7726
  Augmentation therapy: venlafaxine | 14.69
  Monotherapy: Desvenlafaxine: number analyzed (Participants) | 4637
  Monotherapy: Desvenlafaxine | 68.56
  Combination: Desvenlafaxine: number analyzed (Participants) | 4637
  Combination: Desvenlafaxine | 13.48
  Augmentation therapy: desvenlafaxine: number analyzed (Participants) | 4637
  Augmentation therapy: desvenlafaxine | 17.86
  Monotherapy: Mirtazapine: number analyzed (Participants) | 11414
  Monotherapy: Mirtazapine | 71.22
  Combination: Mirtazapine: number analyzed (Participants) | 11414
  Combination: Mirtazapine | 13.01
  Augmentation therapy: mirtazapine: number analyzed (Participants) | 11414
  Augmentation therapy: mirtazapine | 15.92
  Monotherapy: Tianeptine: number analyzed (Participants) | 24536
  Monotherapy: Tianeptine | 65.33
  Combination: Tianeptine: number analyzed (Participants) | 24536
  Combination: Tianeptine | 14.13
  Augmentation therapy: tianeptine: number analyzed (Participants) | 24536
  Augmentation therapy: tianeptine | 13.04
  Monotherapy: Vortioxetine: number analyzed (Participants) | 14504
  Monotherapy: Vortioxetine | 72.53
  Combination: Vortioxetine: number analyzed (Participants) | 14504
  Combination: Vortioxetine | 10.45
  Augmentation therapy: vortioxetine: number analyzed (Participants) | 14504
  Augmentation therapy: vortioxetine | 15.56
  Monotherapy: Bupropion: number analyzed (Participants) | 7698
  Monotherapy: Bupropion | 66.85
  Combination: Bupropion: number analyzed (Participants) | 7698
  Combination: Bupropion | 17.12
  Augmentation therapy: bupropion: number analyzed (Participants) | 7698
  Augmentation therapy: bupropion | 13.78

12. Other Pre Specified Outcome: Drug Utilization Pattern of Participants During 90-180 Days of Treatment
Description: The drug utilization pattern is presented according to the average treatment duration for each antidepressant during the maintenance treatment phases.
Time Frame: From 90 days to 180 days of treatment (data collected and observed retrospectively)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Participants With Antidepressant Therapy
Number analyzed (Participants) | 185842
Days
  Escitalopram: number analyzed (Participants) | 89452
  Escitalopram | 59.05 (27.21)
  Paroxetine: number analyzed (Participants) | 19658
  Paroxetine | 60.50 (26.73)
  Fluoxetine: number analyzed (Participants) | 22100
  Fluoxetine | 56.07 (27.30)
  Sertraline: number analyzed (Participants) | 15984
  Sertraline | 59.58 (26.95)
  Duloxetine: number analyzed (Participants) | 4336
  Duloxetine | 59.25 (27.64)
  Venlafaxine: number analyzed (Participants) | 4065
  Venlafaxine | 61.17 (26.61)
  Desvenlafaxine: number analyzed (Participants) | 2486
  Desvenlafaxine | 63.65 (26.05)
  Mirtazapine: number analyzed (Participants) | 5475
  Mirtazapine | 60.92 (27.17)
  Tianeptine: number analyzed (Participants) | 11339
  Tianeptine | 51.93 (29.53)
  Vortioxetine: number analyzed (Participants) | 7332
  Vortioxetine | 60.91 (26.40)
  Bupropion: number analyzed (Participants) | 3615
  Bupropion | 57.34 (27.18)

ADVERSE EVENTS:
Time Frame: Data for non-serious adverse events and serious adverse events (SAEs) were not collected and evaluated during the study; hence timeframe is not applicable for non-SAEs and SAEs.
Description: This study involved data that existed as structured data and in these data sources, individual participant data could not be retrieved or validated, and it was not possible to link (i.e., identify a potential association between) a particular product and medical event for any individual. The minimum criteria for reporting an adverse event (AE) (i.e., identifiable patient, identifiable reporter, a suspect product, and event) could not be met. Hence, safety data is not reported.
Arm/Group | Participants With Antidepressant Therapy
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT04446039/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT04446039/SAP_001.pdf